CLINICAL TRIAL: NCT06298383
Title: The Effect of Premedication With Trypsin, Bromelain and Rutoside Combination on the Success of IAN Block and Post Endodontic Pain in Patients With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: The Effect of Three Different Medications on Anesthetic Success and Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Egyptian Russian University (Network)
Responsible Party: Principal Investigator, Maha Nasr, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERU1
Record Dates: First submitted 2024-02-19; First posted 2024-03-07 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-06

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Trypsin; Bromelains; Rutin; Diclofenac; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Trypsin, Bromelain and Rutoside (TBR) Group (Experimental): patients will receive Trypsin, Bromelain and Rutoside combination (2 tablets of flamogen a combination of Trypsin 48mg, Bromelain 90mg and Rutoside 100mg) as a single oral dose 1 hour before treatment.
  Interventions: Drug: Trypsin, Bromelain and Rutoside
- NSAIDs Group (Active Comparator): Patients will receive diclofenac potassium (50mg) as a single oral dose 1 hour before treatment.
  Interventions: Drug: Diclofenac Potassium
- Steroid Group (Active Comparator): Patients will receive a single oral dose of a steroid drug (30 mg prednisolone) 1 hour before treatment.
  Interventions: Drug: Prednisolone Oral Tablet
- Placebo group (Placebo Comparator): Patients will receive a single oral dose of placebo (compressed tablets of powdered milk) 1 hour before treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Trypsin, Bromelain and Rutoside — Flamogen is a combination of trypsin 48 mgs, bromelain 90mg and rutoside 100 mg in one tablet that provides an anti inflammatory, anti edematous activity. each patient will receive a single dose of 2 tablets one hour before treatment.
  Other Names: Flamogen
  Arms: Trypsin, Bromelain and Rutoside (TBR) Group
Drug: Diclofenac Potassium — Non-steroidal anti inflammatory drug. cataflam is known for its potent anti inflammatory and analgesic properties. each patient will receive one tablet of cataflam 50 mg 1 hour before treatment.
  Other Names: Cataflam
  Arms: NSAIDs Group
Drug: Prednisolone Oral Tablet — Steroids are potent anti inflammatory drugs, patients are going to receive one tablet of 30 mg solupred one hour before treatment
  Other Names: solupred
  Arms: Steroid Group
Other: Placebo — A tablet of Compacted powdered milk
  Arms: Placebo group

SUMMARY:
Pain is a very important factor in Endodontic treatment, Both intra- and Post-operatively. In case of symptomatic Irreversible pulpitis, a build up of inflammatory mediators makes it very difficult for the operator to reach the desired level of anesthesia in order to deliver a pain free treatment as well as to eliminate or at least reduce post-operative pain incidence and severity. therefore, a number of pre- medications was suggested with variable success rates. Therefore this trial aims at the use of a new category of anti-inflammatory medications which would be less harmful than the standard NSAIDs or steroids.

DETAILED DESCRIPTION:
Background and Rationale

Successful pain management during root canal treatment is crucial for both patients and endodontists. For patients with irreversible pulpitis, achieving adequate pulpal anesthesia during endodontic therapy is a major concern, posing a considerable difficulty from a clinical point of view as an inadequately anesthetized hot tooth with severe pain will not only elevate the patients' apprehension but will also stress the practicing clinician. Inferior alveolar nerve block (IANB) technique is commonly used to achieve pulpal anesthesia in mandibular teeth. Studies reported that the failure ratio of a single IANB block injection of local anesthetic in patients with irreversible pulpitis ranges between 30 and 90 %. Efforts have been made to explain the mechanisms of IANB failure including anatomic variations e.g., cross innervations and accessory innervations, decreased local pH, tachyphylaxis of anesthetic solutions, and activation of nociceptors like tetrodotoxin (TTX) Several clinical studies identified inflammation as a major cause of failure of local anesthesia and an important component of the pathogenesis of hyperalgesia. The use of both steroidal and nonsteroidal anti-inflammatory drugs (NSAIDs) was investigated to improve the success rates of IANB anesthesia, The use of NSAIDs aimed at reducing the chemical inflammatory mediators that activate or sensitize peripheral nociceptors and the related subsequent events involved in pain perception. Because NSAIDs reduce nociceptor activation by decreasing the levels of inflammatory mediators, it is hypothesized that premedication with NSAIDs could affect the success rate of local anesthesia in patients with irreversible pulpitis. Therefore, administration of preoperative NSAIDs to increase the success rate of mandibular molars anesthesia has been studied.

Since both steroidal and NSAID medications are associated with significant side effects, there is a great deal of interest in natural compounds, which have been used for centuries to reduce pain and inflammation. Systemic enzyme therapy refers to the use of proteolytic (hydrolytic) enzymes, also called proteases, which are naturally occurring substances derived from animal or plant sources. Though proteases are mostly known for their role in digestion, they are necessary for some critical processes in the body like protein recycling, immune function, cell division and blood clotting. In our body, these proteases are produced by the stomach and the pancreases; but they are also available in plant and animal sources. The role of proteases is commonly thought of as degradative, but they also contribute to effective immune responses by conveying hormone-like signals and intracellular signal transduction via the specific cell surface receptors. Some of the popular enzymes and their combinations are trypsin-chymotrypsin, bromelain, and papain. Combined with the bioflavonoid rutin (Rutoside), the proteases Trypsin and Bromelain have been extensively investigated as alternatives to conventional therapies for pain and swelling associated with diverse conditions.

The aim of the trial To assess the effect of Trypsin, Bromelain and Rutoside combination versus ibuprofen or dexamethasone or placebo on the anesthetic success of IANB and postoperative pain in patients with symptomatic irreversible pulpitis.

The null hypothesis tested is " In patients with symptomatic irreversible pulpitis in their mandibular molars, there is no difference between Trypsin, Bromelain and Rutoside combination or ibuprofen or dexamethasone or placebo on anesthetic success and post-operative pain after endodontic treatment."

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic irreversible pulpitis.
* Patients with active pain (moderate-to-severe) in mandibular molars.
* Males and females.
* Patient with the ability to understand and use pain scales.
* Patient who accepts to enroll to the study

Exclusion Criteria:

* Patients' allergies or any other contraindication to any of the used medications or mepivacaine.
* Pregnant and lactating females.
* Patients have been taking pain medication 12 hours earlier.
* Patient has more than one symptomatic mandibular tooth in the same quadrant.
* Patients with periradicular pathosis and/or radiolucency other than widened periodontal ligaments.
* Patients with contributory medical history (ASA>II).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Success of Anesthesia | through study completion "an average of 1 year"
  Success of Inferior alveolar Nerve block anesthesia will be measured by recording the patient's pain severity before and after anesthesia administration as well as during endodontic procedures. each patient will record his/her pain on a "Numerical Rating Scale" (NRS), the NRS is an eleven point scale anchored at both ends by zero representing no pain and 10 representing pain as bad as it could be.
Post-operative pain | through study completion "an average of 1 year"
  postoperative pain as recorded by the patient after completion of treatment in on visit.
  patient will receive a pain diary to record their postoperative pain incidence and severity at 6, 12, 24, 72 hours and 7 days after endodontic treatment.
  Each patient will record his/her pain on a "Numerical Rating Scale" (NRS), the NRS is an eleven point scale anchored at both ends by zero representing no pain and 10 representing pain as bad as it could be.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Nasr, Principal Investigator — Egyptian Russian University
Locations (2):
- Egypt (2):
  - Faculty of Oral and Dental Medicine, Egyptian Russian University, Cairo, Cairo Governorate
  - Faculty of Dentistry, Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No